CLINICAL TRIAL: NCT00946855
Title: Laboratory Values in Elite Soccer Players
Brief Title: Effect of Elite Soccer Training on Routine Laboratory Parameters
Acronym: SOCCERLAB
Status: Completed | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Prof. Dr. med. Tim Meyer, Institute of Sports and Preventive Medicine, University of Saarland, Campus Bldg. B 8-2, 66123 Saarbrücken, Germany
Other Study IDs: Soccer laboratory values
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2009-07-27 (Estimated); Status verified 2009-07

CONDITIONS: Stress
Keywords: soccer; laboratory; reference; exercise; variability; season; elite athletes; Define reference blood parameters in elite athletes
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — iced serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- soccer players: players of the first two German soccer leagues

SUMMARY:
Repeated blood sampling within a regular soccer season of German first league clubs shall serve to define soccer-specific reference values for routine parameters determined from venous blood. It was hypothesized that only for a minor number of parameters common reference values will have to be adapted for soccer players during their competitive season.

DETAILED DESCRIPTION:
It is often difficult to discern exercise-induced changes in laboratory parameters from pathological changes in elite athletes during the regular training process. This is particularly true in soccer players who compete more often than many other athletes. Therefore, soccer players of the first two German soccer leagues (all professional athletes) are recruited for repeated blood sampling during the season (4 sampling times, one of them immediately before training commences in the summer, the other ones in October/November, February/March, and April/May). Among other standardizing requirements, it is mandatory that precisely one training session (not zero, not two, no competition) takes place the day before sampling. Several confounders for the interpretation of laboratory results are verified by means of a questionnaire. Phases of high competitive stress are compared with those of low stress. The course of the parameters as well as confidence intervals for given times during the season are of main interest.

ELIGIBILITY:
Inclusion Criteria:

* being employed as player by a club of the first two German soccer leagues
* healthy

Exclusion Criteria:

* chronic disease interfering with one or more of the determined parameters

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: soccer players of the first two German professional soccer leagues
Sampling Method: Non-Probability Sample
Enrollment: 467 (Actual)
Dates: Start 2008-08; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
complete blood count | August 2008 until May 2009

SECONDARY OUTCOMES:
numerous serum parameters from venous blood | August 2008 until May 2009

CONTACTS AND LOCATIONS:
Overall Officials: Tim Meyer, MD, PhD, Principal Investigator — Institute of Sports and Preventive Medicine, University of Saarland, Campus, Bldg. B 8-2, 66123 Saarbrücken, Germany
Locations (1):
- Institute of Sports and Preventive Medicine, University of Saarland, Campus, Bldg. B 8-2,, Saarbrücken, Saarland, Germany

REFERENCES:
- [Derived] Breitbart P, Meister S, Meyer T, Gartner BC. Incidence and Prevalence of Borrelia burgdorferi Antibodies in Male Professional Football Players. Clin J Sport Med. 2021 Jul 1;31(4):e200-e206. doi: 10.1097/JSM.0000000000000758. PMID 31241490
- [Derived] Meyer T, Meister S. Routine blood parameters in elite soccer players. Int J Sports Med. 2011 Nov;32(11):875-81. doi: 10.1055/s-0031-1280776. Epub 2011 Oct 21. PMID 22020850
- See also: Homepage of study center — http://www.sportmedizin-saarbruecken.de